CLINICAL TRIAL: NCT04780373
Title: Identification of a Clinical Score to Support the Clinician in Phase 2 of Covid-19
Brief Title: Prognostic Score in Covid-19
Status: Completed | Type: Observational
Sponsor: University of L'Aquila (Other)
Responsible Party: Principal Investigator, Clara Balsano, Full Professor, University of L'Aquila
Other Study IDs: prot. N. 71726
Record Dates: First submitted 2021-01-22; First posted 2021-03-03 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Covid19 Prognostic Parameters
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Development cohort
  Interventions: Other: data collection
- Validation cohort
  Interventions: Other: data collection

INTERVENTIONS:
Other: data collection — clinical data collection

SUMMARY:
The aim of the study is to define the clinical and biochemical parameters that characterize COVID-19 patients with a negative prognostic evolution. Our clinical score will be capable to recognize patient with favorable prognosis or patient with poor prognosis by statistical data analysis.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 and symptomatic and positive for COVID-19 by polymerase chain reaction assay for rhino-pharingeal swab

Exclusion Criteria:

* Under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Italian Caucasian Patients ≥ 18 years old SARS-CoV-2 infection confirmed by PCR
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Data collection of clinical and demographical parameters of patients affected by COVID-19 | 8 months
  Data about sex, age, symptom start date, vital parameters, comorbidity, symptoms, hematochemicals blood tests, therapy, oxygen support, radiology, condition evaluation will be manual collected.

SECONDARY OUTCOMES:
Application of statistical analysis on data of patients affected by COVID-19 | 2 months
  The collected data will be analyzed through descriptive statistics analysis, ROC curves, regression analysis, and Machine Learning techniques to predict the prognosis of patients affected by COVID-19.

CONTACTS AND LOCATIONS:
Locations (1):
- University of L'Aquila, L’Aquila, Italy

REFERENCES:
- [Derived] Sinatti G, Santini SJ, Tarantino G, Picchi G, Cosimini B, Ranfone F, Casano N, Zingaropoli MA, Iapadre N, Bianconi S, Armiento A, Carducci P, Ciardi MR, Mastroianni CM, Grimaldi A, Balsano C. PaO2/FiO2 ratio forecasts COVID-19 patients' outcome regardless of age: a cross-sectional, monocentric study. Intern Emerg Med. 2022 Apr;17(3):665-673. doi: 10.1007/s11739-021-02840-7. Epub 2021 Oct 12. PMID 34637082